CLINICAL TRIAL: NCT02108704
Title: Helicobacter Pylori Eradication in Parkinson's Disease: A Double-blind Randomised Placebo Controlled Trial
Brief Title: Helicobacter Pylori Eradication Study in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HPPD
Record Dates: First submitted 2014-04-04; First posted 2014-04-09 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Parkinson's Disease; Helicobacter Pylori Infection
Keywords: Parkinson's Disease; Helicobacter pylori infection
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Helicobacter pylori eradication therapy (Active Comparator): Amoxycillin 1gm twice a day (BD) Clarithromycin 500mg BD Omeprazole 20mg BD
  Interventions: Drug: Helicobacter pylori eradication therapy
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Helicobacter pylori eradication therapy
  Arms: Helicobacter pylori eradication therapy
Drug: Placebo
  Arms: Placebo

SUMMARY:
It has been hypothesized, based on epidemiological observations, that Helicobacter pylori (HP) infection may play a role in the pathogenesis of Parkinson's Disease (PD). Previous studies have also shown that HP eradication therapy may result in improvements in levodopa pharmacokinetics and motor fluctuations. This study aims to examine the effects of HP eradication, using a double-blind randomized placebo-controlled trial design in a relatively large cohort of patients. Outcomes of interest include motor function, gastrointestinal symptoms and health-related quality of life. The investigators hypothesize that HP eradication will lead to improvements in motor function. The primary outcome of interest is the "ON"-medication Unified PD Rating Scale (UPDRS) Part III score at 3 months. Secondary outcomes include Purdue Pegboard Score, Timed Test of Gait, Dyskinesia and Bradykinesia scores measured by Parkinson's Kinetigraph (PKG), Leeds Dyspepsia Questionnaire (LDQ), Parkinson's Disease Questionnaire (PDQ-39), UPDRS Part I, Part II and Part IV; and Montreal Cognitive Assessment (MOCA).

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years
2. Provision of written informed consent
3. Clinical diagnosis of Parkinson's Disease (PD) assigned by a consultant neurologist

Exclusion Criteria:

1. History of previous gastric or major abdominal/pelvic surgery
2. History of previous eradication therapy for Helicobacter pylori
3. Antibiotic use in the preceding four weeks or use of anti-acid/prokinetics/laxatives in the preceding one week prior to breath test
4. Recent initiation of dopaminergic medications (within the last three months) or recent adjustment of dopaminergic medications (within the last one month)
5. History of functional neurosurgery for PD
6. No concomitant neurologic disease except PD
7. Medical condition that prevents reliable completion of questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
"On-medication" MDS-UPDRS Part III score | at 3 months after randomisation

SECONDARY OUTCOMES:
"On-medication" UPDRS Part III score | at 1 year post randomisation
"On-medication" Pegboard Score | at 3 months and 1 year post randomisation
"On-medication" Timed Gait Score | at 3 months and 1 year post randomisation
Parkinson's Kinetigraph (PKG) Bradykinesia and Dyskinesia Scores | at 3 months and 1 year post randomisation
UPDRS Part IV | at 3 months and 1 year post randomisation
UPDRS Part II | at 3 months and 1 year post randomisation
UPDRS Part I | at 3 months and 1 year post randomisation
Montreal Cognitive Assessment Score | at 3 months and 1 year post randomisation
Leeds Dyspepsia Questionnaire | at 3 months and 1 year post randomisation
Parkinson Disease Questionnaire (PDQ-39) | at 3 months and 1 year post randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Ai Huey Tan, MD,MRCP(UK), Principal Investigator — University of Malaya
Locations (1):
- University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia